CLINICAL TRIAL: NCT02064712
Title: Determining an Optimal Weaning Method of Nasal Continuous Positive Airway Pressure in Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCPAPwean
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Infant, Newborn; Infant, Premature
Keywords: Continuous Positive Airway Pressure
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low CPAP Wean (Active Comparator): NCPAP weaned to 5cm H2O for minimum of 24h, and if the neonate remains clinically stable as defined, wean in 1cm increments to 3cm H2O for minimum of 24h, at which time move to room air or 1L/min nasal cannula if supplemental O2 is required.
  Interventions: Other: Low CPAP Wean
- High CPAP Wean (Active Comparator): NCPAP weaned to 5cm H2O for a minimum of 24h, and if the neonate remains clinically stable, move to room air or 1L/min nasal cannula if supplemental O2 is required.
  Interventions: Other: High CPAP Wean

INTERVENTIONS:
Other: Low CPAP Wean — Infants receive NCPAP by Hudson nasal prongs.
  Arms: Low CPAP Wean
Other: High CPAP Wean — Infants receive NCPAP by Hudson nasal prongs.
  Arms: High CPAP Wean

SUMMARY:
The purpose of this study is to determine an optimal strategy to wean nasal continuous positive airway pressure (NCPAP) in preterm babies. The investigators hypothesize that babies that are taken off NCPAP at lower settings will need fewer total days on NCPAP than those babies taken off at higher settings.

DETAILED DESCRIPTION:
This is a prospective randomized control trial to investigate an optimal method for discontinuing NCPAP therapy in preterm neonates. Neonates ≤32 weeks gestational age (GA) who require NCPAP in the delivery room or following extubation and are delivered in or transferred to Parkland Hospital Neonatal Intensive Care Unit (NICU) will be enrolled. The study team will approach the parents for verbal consent once neonates are stable on mechanical ventilation with a goal of extubation to NCPAP or once they are placed on initial NCPAP therapy. Neonates will be randomized to the high or low NCPAP arms and managed by their primary care team until they meet stability criteria as defined for a minimum of 12 hours. At that time they will be removed from NCPAP using two approaches: Group 1 will be decreased to 5cm H2O by the primary care team at which time NCPAP is removed if the neonate is clinically stable and the neonate placed in room air or on low-flow nasal cannula at ≤1L/min; Group 2 will be gradually weaned to a NCPAP of 3cm H2O at which time NCPAP is removed if the neonate is clinically stable for the prior 24 hours and the neonate placed in room air or on low-flow nasal cannula. Failure criteria will consist of clinical signs and laboratory results demonstrating the need for escalation of support, e.g., increasing apnea of prematurity (AOP) or need for increasing O2 supplementation. When a neonate has been stable for 5 days off NCPAP, they will complete the intervention arm of the study. All neonates will be followed until discharge, at which time the primary outcomes, e.g., days on NCPAP, duration of hospitalization and need for O2, will be determined for each group and compared. The calculated total sample size will require 238 neonates; i.e., 113 neonates per arm with a 5% drop-out rate will give a power of 0.80 and alpha value of 0.05 to detect a 25% difference in NCPAP days.

Stability Criteria:

1. NCPAP 5cm H2O
2. Supplemental oxygen <25% and not increasing
3. Respiratory rate ≤60 b/min
4. No significant respiratory distress, e.g., retractions, dyspnea
5. <3 episodes of apnea (>20 seconds) with bradycardia (<100 beats/min), and/or desaturations (<88%) within 1h or <5 episodes in prior 12h
6. Average oxygen saturation >87% with stable inspired O2
7. Tolerate time off NCPAP during routine care procedures
8. Neonates <27 wks GA must be ≥10d postnatal before weaning

Failure Criteria:

1. Occurrence of ≥3 apneas and/or bradycardia and/or desaturations within 1h or >4 episodes in a 12h period
2. Increasing need for supplemental O2 >30% to maintain O2 saturation >87%
3. Increase in the PaCO2 >65 mmHg
4. Increased work of breathing with respiratory rate >75 b/min for >2h
5. AOP requiring resuscitation
6. Initiation of nasal intermittent positive pressure ventilation (NIPPV) for respiratory support

ELIGIBILITY:
Inclusion Criteria:

* Neonates ≤32wks GA requiring NCPAP in the delivery room or NICU for increasing respiratory distress or post-extubation from mechanical ventilation.

Exclusion Criteria:

* Neonates requiring NCPAP for less than 48 hours
* Congenital anomalies
* Need for surgery
* Transfer to a different facility
* Grade 3-4 intraventricular hemorrhage

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 226 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Total days of NCPAP | Until hospital discharge or 1 year of life
  Total number of days of CPAP therapy during the hospital stay

SECONDARY OUTCOMES:
Length of hospital stay | Until hospital discharge or 1 year of life
  Number of days spent prior to being discharged from the hospital
Duration of oxygen supplementation | Until hospital discharge or 1 year of life
  Number of days

CONTACTS AND LOCATIONS:
Overall Officials: Venkat Kakkilaya, MD, Principal Investigator — UT Southwestern
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

REFERENCES:
- [Derived] Kakkilaya V, Tang A, Wagner S, Ridpath J, Ibrahim J, Brown LS, Rosenfeld CR. Discontinuing Nasal Continuous Positive Airway Pressure in Infants </=32 Weeks of Gestational Age: A Randomized Control Trial. J Pediatr. 2021 Mar;230:93-99.e3. doi: 10.1016/j.jpeds.2020.10.045. Epub 2020 Oct 28. PMID 33127365